CLINICAL TRIAL: NCT01787682
Title: Metabolic and Functional Changes in Relation to Nutritional Status in Chronic Heart Failure and Chronic Obstructive Pulmonary Disorder
Brief Title: Nutritional and Functional Changes in Heart Failure and COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-0503
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Chronic Heart Failure; Chronic Obstructive Pulmonary Disorder
Keywords: CHF; Protein digestion; Fat digestion; Gut function; Glucose absorption; Muscle function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Boost High Protein (Experimental): Boost high protein with added spirulina
  Interventions: Dietary Supplement: BOOST High Protein

INTERVENTIONS:
Dietary Supplement: BOOST High Protein

SUMMARY:
Weight loss commonly occurs in patients with chronic heart failure (CHF) and chronic obstructive pulmonary disorder (COPD), negatively influencing their quality of life, treatment response and survival. Loss of muscle protein is generally a central component of weight loss in CHF and COPD patients but patients also have reductions in fat mass and bone density, independent of the severity of the disease state. The purpose of this cross-sectional study is to provide detailed insight in disease related gut function by obtaining information on gut permeability, digestion and absorption of glucose, fat and protein in CHF and COPD patients compared to matched healthy controls. This will provide required information that is necessary to implement new strategies to develop optimal nutritional regimen in CHF and COPD. The hypothesis is that CHF and COPD are related to decreased gut function and absorption, leading to decreased anabolic response. Second, this decreased nutritional status is linked to reduced muscle functioning and possibly decreased cognition. In addition, we will examine the effect of aging on by comparing gut function digestion and absorption of the CHF and COPD aged matched healthy controls to a group of young healthy subjects.

DETAILED DESCRIPTION:
This study involves one test day of approximately 7-8 hours. On this test day subjects will ingest a sugar drink to assess gut permeability and gut function, and a protein meal to measure digestion/absorption and the anabolic response to food intake. Subjects will also receive a mixture of amino acids that are made a little heavier than normal, called stable isotopes. This stable isotopes is used to investigate protein behavior in the body (protein kinetics). Blood (100-120 ml in total) and urine samples will be collected over 7 hours.

ELIGIBILITY:
Inclusion criteria CHF subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 7 hours
* Diagnosis of Chronic Heart Failure; under regular care by cardiologist
* NYHA class II-IV
* Reduced ejection fraction (<45%) assessed in the past 2 years
* Clinically stable condition; no hospitalization 4 weeks preceding first study day
* Willingness and ability to comply with the protocol

Inclusion criteria COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 8 hours
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol

Inclusion criteria healthy control subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 45 years or older (older control group)
* Age between 20-30 years old (young group)
* Ability to lay in supine or elevated position for 7 hours
* No diagnosis of CHF
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Body mass index >40 kg/m2 (healthy subjects only)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Use of protein or amino acid containing nutritional supplements within 5 days of first study day
* Current use of long-term oral corticosteroids (CHF only)
* Use of short course of oral corticosteroids within 4 weeks preceding first study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-12; Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Net whole-body protein synthesis | 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 min post-meal
  change in whole-body protein synthesis rate after intake of meal

SECONDARY OUTCOMES:
Citrulline Rate of appearance | Postabsorptive state during 2 hours
  plasma enrichment of citrulline
Glucose absorption | 7 hours
  Recovery of 3-O-Methyl-D-glucose in the urine.
Gut permeability | 7 hours
  recovery of rhamnose/lactulose in urine
Skeletal and respiratory muscle strength | 1 day
  Difference in leg strength and fatigue, handgrip strength and fatigue, and inspiratory and expiratory pressure between heart failure patients and healthy controls.
Cognitive function | 1 day
  Outcome of neuro-psychological tests in heart failure patients and healthy controls in relation to the tryptophan metabolism
Fatty acid digestion after feeding | 0,15,30,45,60,75,90,105,120,150,180,210 min post-meal
  Enrichment in palmitic acid and tripalmitin fatty acids in plasma
Protein digestion after feeding | 0,15,30,45,60,75,90,105,120,150,180,210, min post-meal
  Ratio enrichment free phenylalanine vs phenylalanine from protein spirulina
Arginine turnover rate | postabsorptive state during 3 hours
  Arginine enrichment in plasma
Whole body collagen breakdown rate | Postabsorptive state during 3 hours
  Hydroxyproline enrichment in plasma
Tryptophan turnover rate | Postabsorptive state during 3 hours
  Tryptophan enrichment in plasma
Insulin response to feeding | during 3 hours after feeding
  Acute change from postabsorptive state after intake of meal
Fat-free mass | postabsorptive state during 15 min
  Characteristics of study subjects
Myofibrillar protein breakdown rate | 0,15,30,45,60,75,90,105,120,150,180,210 min post-meal
  3methylhistidine enrichment in plasma
Glycine rate of appearance | Postabsorptive state during 3 hours
  glycine enrichment in plasma
Taurine turnover rate | postabsorptive state during 3 hours
  enrichment of taurine in

CONTACTS AND LOCATIONS:
Overall Officials: Marielle PKJ Engelen, PhD, Principal Investigator — Texas A&M Univeristy
Locations (1):
- Texas A&M University, College Station, Texas, United States

REFERENCES:
- [Derived] Deutz LN, Wierzchowska-McNew RA, Deutz NE, Engelen MP. Reduced plasma glycine concentration in healthy and chronically diseased older adults: a marker of visceral adiposity? Am J Clin Nutr. 2024 Jun;119(6):1455-1464. doi: 10.1016/j.ajcnut.2024.04.008. Epub 2024 Apr 12. PMID 38616018
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951
- [Derived] Wierzchowska-McNew RA, Engelen MPKJ, Thaden JJ, Ten Have GAM, Deutz NEP. Obesity- and sex-related metabolism of arginine and nitric oxide in adults. Am J Clin Nutr. 2022 Dec 19;116(6):1610-1620. doi: 10.1093/ajcn/nqac277. PMID 36166849
- [Derived] Pinson MR, Deutz NEP, Harrykissoon R, Zachria AJ, Engelen MPKJ. Disturbances in branched-chain amino acid profile and poor daily functioning in mildly depressed chronic obstructive pulmonary disease patients. BMC Pulm Med. 2021 Nov 7;21(1):351. doi: 10.1186/s12890-021-01719-9. PMID 34743729
- [Derived] Engelen MPKJ, Jonker R, Thaden JJ, Ten Have GAM, Jeon MS, Dasarathy S, Deutz NEP. Comprehensive metabolic flux analysis to explain skeletal muscle weakness in COPD. Clin Nutr. 2020 Oct;39(10):3056-3065. doi: 10.1016/j.clnu.2020.01.010. Epub 2020 Jan 29. PMID 32035752
- [Derived] Deutz NEP, Thaden JJ, Ten Have GAM, Walker DK, Engelen MPKJ. Metabolic phenotyping using kinetic measurements in young and older healthy adults. Metabolism. 2018 Jan;78:167-178. doi: 10.1016/j.metabol.2017.09.015. Epub 2017 Oct 3. PMID 28986165